CLINICAL TRIAL: NCT07087951
Title: Development and Validation of an Innovative Gamma Auditory Stimulation System for Older Adults With Cognitive Decline: A Randomized, Double-blind, Placebo-controlled Study (Study 1)
Brief Title: Efficacy of Gamma Auditory Stimulation for Cognitive Decline in Older Adults (Study 1)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202402079B0A3
Record Dates: First submitted 2025-07-07; First posted 2025-07-28 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-04

CONDITIONS: EEG Brain Oscillations; Alzheimer's Disease (AD) and Related Disorders; Cognitive Dysfunction
Keywords: endogenous gamma; EEG rhythms; resting-state EEG (rs-EEG); Alzheimer's disease (AD); Cognitive function; auditory stimulation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40Hz music group (Experimental): The 40Hz music is combined with 40Hz sound and music.
  Interventions: Device: Gamma auditory stimulation device (active setting)
- Non-40Hz music group (Sham Comparator): The non-40Hz music is combined with non-40Hz sound and music.
  Interventions: Device: Gamma auditory stimulation device (sham setting)

INTERVENTIONS:
Device: Gamma auditory stimulation device (active setting) — Participants will receive auditory stimulation using the gamma auditory stimulation device (active setting) for 1 hour per day, 5 days a week, over 12 weeks, for a total of 60 hours.
  Arms: 40Hz music group
Device: Gamma auditory stimulation device (sham setting) — Participants will receive auditory stimulation using the gamma auditory stimulation device (sham setting) for 1 hour per day, 5 days a week, over 12 weeks, for a total of 60 hours.
  Arms: Non-40Hz music group

SUMMARY:
Animal studies have shown that 40 Hz auditory stimulation alone can improve spatial memory and reduce Aβ deposition. However, human studies using 40 Hz auditory stimulation alone remain limited. Therefore, this study will use a randomized, double-blind, placebo-controlled design to investigate the effects of 40 Hz auditory stimulation on cognitive function, EEG activity, sleep quality, and quality of life in older adults with mild cognitive impairment (MCI) or mild dementia.

DETAILED DESCRIPTION:
Amyloid-beta (Aβ) aggregation and hyperphosphorylated tau protein tangles are widely recognized as the main pathological features of Alzheimer's disease (AD). Numerous domestic and international studies have demonstrated that 40 Hz gamma visual stimulation can effectively enhance 40 Hz gamma neural oscillations in healthy adults and older adults, improve cognitive performance and memory function in older adults and individuals with AD, and has shown good safety with no severe adverse effects.

Nevertheless, there are still several limitations to using 40 Hz visual stimulation as an intervention. Extended exposure to light sources may cause discomfort, affecting participants' willingness to continue. Prolonged light exposure may also increase the risk of seizures in photosensitive individuals. In addition, participants are required to actively fixate on the light source, which may reduce intervention adherence. Most importantly, the ecological validity of light-based stimulation remains low. Many studies require participants to gaze at light for at least five minutes or more, and daily sessions of up to an hour over several months are challenging to implement in daily life. To address these limitations, this project proposes using 40 Hz auditory stimulation as a more practical and sustainable intervention.

Moreover, animal studies have confirmed that 40 Hz auditory stimulation alone can improve spatial memory and reduce Aβ deposition. However, evidence on the independent application of 40 Hz auditory stimulation in humans remains limited. Therefore, this project will adopt a randomized, double-blind, placebo-controlled design to investigate the effects of 40 Hz auditory stimulation on cognitive function, EEG activity, sleep quality, and quality of life in older adults with mild cognitive impairment (MCI) or mild dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 60 years old.
2. MMSE≤ 24
3. CDR scores of 0.5 and 1
4. Voluntary to sign the Informed Consent Form.

Exclusion Criteria:

1. Diagnosis of other psychiatric or neurological disorders
2. Drug or alcohol addictions.
3. Serious heart, liver or kidney disorders, and visual, auditory or motor impairments interfering with neuropsychological tests.
4. History of clinical stroke, major depressive disorder or dysthymic disorder according to the DSM-5.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in neurophysiological function. | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  The changes of power spectral density (PSD) and functional connectivity (FC) at each frequency band will be analyzed by EEG data from each subject.

SECONDARY OUTCOMES:
Change score of the Chinese version Verbal Learning Test (CVVLT). | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  A nine-item of CVVLT (total recall, delayed recall) will be applied to measure the participant's memory ability, with a higher score indicating better performance.
Change score of the WMS-III logical memory test | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  WMS-III logical memory test (immediate recall, delayed recall) will be applied to measure the participant's memory ability. The maximum score is 25 for each recall trial, with a higher score indicating better performance
Change score of the Taylor Complex Figure Test (TCFT). | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  TCFT (immediate recall, delayed recall) will be applied to measure the participant's memory ability. The maximum score is 36 for each recall trial, with a higher score indicating better performance
Change score of the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  A neuropsychological test used to assess cognitive impairment, particularly in the context of Alzheimer's disease. The ADAS-Cog typically has a total score ranging from 0 to 70, with higher scores indicating greater cognitive impairment.
Change score of the Cognitive Abilities Screening Instrument (CASI). | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  CASI will be applied to measure the participant's general cognitive ability. The range of score is 0 to 100, with a higher score indicating better performance.
Change score of the category Verbal Fluency Test (VFT). | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  The category VFT will be applied to measure the participant's language and executive function, with a higher score indicates better performance.
Performance changes of the Trail Making Test Form A/B (TMT-A/B) | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  TMT-A/B will be applied to measure participant's attention and executive function. The number of seconds to complete each trial and the number of errors would be recorded, with a higher value indicating greater impairment.
Performance changes of the Digit Span Test | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  This is a widely used neuropsychological assessment that measures attention (Digit Span Forward), and working memory (Digit Span Backward). If the participant correctly repeats the digit sequence, the number of digits in the next sequence will increase. The test will be terminated after a set number of errors.
Change score of the neuropsychiatric Inventory (NPI) | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  It evaluates 12 neuropsychiatric domains. For each symptom, the NPI assesses both its frequency (how often it occurs) and severity (how intense it is). A higher score indicates more severe symptom.
Change score of the Geriatric Depression Scale -short form (GDS-S) | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  This tool consists of 15 yes-or-no questions and is commonly used to assess depression in older adults. A higher score indicates more severe depression.
Change score of the Pittsburgh Sleep Quality Index (PSQI) | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  It used to comprehensively assess participants' sleep quality over the past month with 19 questions. Each component is scored from 0 to 3, with higher scores indicating greater sleep problems. The total PSQI score, a sum of all component scores, will range from 0 to 21, where a score above 5 indicates poor sleep quality.
Change score of the 5-level EuroQol-5 Dimension (EQ-5D-5L) | baseline (T1), through intervention completion, an average of 3 month (T2), three-month after intervention completion (T3)
  It used to assess an individual's quality of life with five questions and each dimension has five levels of severity. Additionally, the EQ-5D-5L includes a Visual Analog Scale, where respondents rate their overall health on a scale from 0 (the worst imaginable health) to 100 (the best imaginable health).
Safety/Adverse events outcome measure | Throughout the three-months intervention
  Adverse events, such as fatigue, headache, dizziness, dazzling, ear pain, and others, will be recorded using a 6-point Likert scale ranging from 'not at all' to 'extremely uncomfortable' (0 = not at all, 1 = minimal discomfort, 2 = mild discomfort, 3 = tolerable, 4 = severe discomfort, 5 = extreme discomfort).
  Participants will report adverse events (such as fatigue, headache, dizziness, dazzling, ocular pain, and others) using a 6-point Likert scale ranging from 'not at all' to 'extremely uncomfortable' after each light stimulation session.
Device feasibility outcome measure | Throughout the three-months intervention
  Participants will answer a device feasibility questionnaire, include "how is the usability of the device", "How is your satisfaction of the user interface " ...etc. We will use a 6-point Likert scale ranging from 'not at all' to 'extremely good'.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: No